CLINICAL TRIAL: NCT02846441
Title: Interstage Assessment of Remnant Liver Function in ALPPS: Can SPECT Hepatobiliary Scintigraphy Provide Any Additional Value in Predicting Risk of Posthepatectomy Liver Failure?
Brief Title: Interstage Assessment of Remnant Liver Function in ALPPS
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, eduardo de santibanes, MD, PhD, Hospital Italiano de Buenos Aires
Other Study IDs: 2900
Record Dates: First submitted 2016-07-22; First posted 2016-07-27 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Liver Failure
Keywords: posthepatectomy liver failure; ALPPS; hepatobiliary scintigraphy; SPECT; mebrofenin
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: hepatobiliary scintigraphy — 99mTc-mebrofenin hepatobiliary scintigraphy with single photon emission computed tomography (SPECT)
  Other Names: spect

SUMMARY:
Post-hepatectomy liver failure is one of the most feared complications by hepatic surgeons. When size of the future liver remnant (FLR) is regarded to be not sufficient to sustain post-hepatectomy liver function, techniques as preoperative portal vein embolization or two-stage hepatectomy/associating liver partition and portal vein ligation (ALPPS) can be performed. ALPPS induces rapid and extensive hypertrophy by portal vein ligation and in situ liver splitting. To date, feasibility of the second stage of ALPPS has been assessed only on the basis of standardized future liver remnant or future liver remnant on body weight. However, decrease of liver function between stages, measured by means of laboratory parameters, has been demonstrated to be associated with higher 90-day mortality, regardless of FLR volume. In other words, this volumetric increase may not reflect the increase of liver function.

DETAILED DESCRIPTION:
The aim of this study is to determine the predictive value of hepatobiliary scintigraphy with 99mTc-mebrofenin between stages in ALPPS, in assessing risk of postoperative liver failure and liver failure-related mortality after completion of stage 2.

ELIGIBILITY:
Inclusion Criteria:

* Hepatobiliary scintigraphy performed between stages in patients submitted to ALPPS surgery
* Aged ≥18

Exclusion Criteria:

* Known allergy to Hida derivatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients submitted to ALPPS surgery at the Hospital Italiano between 2011 and 2016.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
posthepatectomy liver failure | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: eduardo de santibanes, MD, PhD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ekman M, Fjalling M, Holmberg S, Person H. IODIDA clearance rate: a method for measuring hepatocyte uptake function. Transplant Proc. 1992 Feb;24(1):387-8. No abstract available. PMID 1539327
- [Background] de Graaf W, van Lienden KP, Dinant S, Roelofs JJ, Busch OR, Gouma DJ, Bennink RJ, van Gulik TM. Assessment of future remnant liver function using hepatobiliary scintigraphy in patients undergoing major liver resection. J Gastrointest Surg. 2010 Feb;14(2):369-78. doi: 10.1007/s11605-009-1085-2. PMID 19937195
- [Background] de Graaf W, van Lienden KP, van Gulik TM, Bennink RJ. (99m)Tc-mebrofenin hepatobiliary scintigraphy with SPECT for the assessment of hepatic function and liver functional volume before partial hepatectomy. J Nucl Med. 2010 Feb;51(2):229-36. doi: 10.2967/jnumed.109.069724. Epub 2010 Jan 15. PMID 20080899
- [Background] Schadde E, Raptis DA, Schnitzbauer AA, Ardiles V, Tschuor C, Lesurtel M, Abdalla EK, Hernandez-Alejandro R, Jovine E, Machado M, Malago M, Robles-Campos R, Petrowsky H, Santibanes ED, Clavien PA. Prediction of Mortality After ALPPS Stage-1: An Analysis of 320 Patients From the International ALPPS Registry. Ann Surg. 2015 Nov;262(5):780-5; discussion 785-6. doi: 10.1097/SLA.0000000000001450. PMID 26583666
- [Background] Rahbari NN, Garden OJ, Padbury R, Brooke-Smith M, Crawford M, Adam R, Koch M, Makuuchi M, Dematteo RP, Christophi C, Banting S, Usatoff V, Nagino M, Maddern G, Hugh TJ, Vauthey JN, Greig P, Rees M, Yokoyama Y, Fan ST, Nimura Y, Figueras J, Capussotti L, Buchler MW, Weitz J. Posthepatectomy liver failure: a definition and grading by the International Study Group of Liver Surgery (ISGLS). Surgery. 2011 May;149(5):713-24. doi: 10.1016/j.surg.2010.10.001. Epub 2011 Jan 14. PMID 21236455
- [Background] Schnitzbauer AA, Lang SA, Goessmann H, Nadalin S, Baumgart J, Farkas SA, Fichtner-Feigl S, Lorf T, Goralcyk A, Horbelt R, Kroemer A, Loss M, Rummele P, Scherer MN, Padberg W, Konigsrainer A, Lang H, Obed A, Schlitt HJ. Right portal vein ligation combined with in situ splitting induces rapid left lateral liver lobe hypertrophy enabling 2-staged extended right hepatic resection in small-for-size settings. Ann Surg. 2012 Mar;255(3):405-14. doi: 10.1097/SLA.0b013e31824856f5. PMID 22330038